CLINICAL TRIAL: NCT02858570
Title: Immunogenicity, Reactogenicity and Safety Assessment of the Meningococcal Serogroup C Vaccine Produced by Bio-Manguinhos / FIOCRUZ in Infants, Children and Adolescents
Brief Title: Conjugate Vaccine Against Meningococcus C a Brazilian Project
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ASCLIN 001/2016
Record Dates: First submitted 2016-07-26; First posted 2016-08-08 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Serogroup C Meningococcal Meningitis
Keywords: Meningococcal Vaccines; Immunogenicity, Reactogenicity and Safety of Vaccine
MeSH Terms: conditions — Meningitis, Meningococcal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MenCC-BIO Vaccine (Experimental): Vaccine against meningococcus serogroup C conjugated to tetanus toxoid produced by Bio-Manguinhos / FIOCRUZ (MenCC-Bio). Stratum I - 11-19 years; Stratum II - 1 to 10; Stratum III - less than 1 year old)For the age groups I and II are applied 2 doses ideal interval of 6 months between them. In stratum III, are recommended 3 doses of the vaccine, at ages 3, 5 and 12 months of age, according to calendar of the National Immunization Program.
  Interventions: Biological: MenCC-BIO Vaccine
- combined - CRM197 (Active Comparator): Adsorbed vaccine meningococcal C (combined - CRM197) produced by the Foundation Ezequiel Dias (FUNED). Stratum I - 11-19 years; Stratum II - 1 to 10; Stratum III - less than 1 year old). For the age groups I and II are applied 2 doses ideal interval of 6 months between them. In stratum III, are recommended 3 doses of the vaccine, at ages 3, 5 and 12 months of age, according to calendar of the National Immunization Program.
  Interventions: Biological: Combined - CRM197

INTERVENTIONS:
Biological: MenCC-BIO Vaccine — The Bio-MenCC vaccine is composed of serogroup C meningococcal polysaccharide conjugated to tetanus toxoid as the carrier protein, with 10 microgram of capsular polysaccharide of group C, 10-20 microgram of tetanus toxoid per dose and aluminum hydroxide at a concentration of 1 milligram dose (0.35 milligram Al3 +) with phosphate buffered saline as diluent. The vaccine is lyophilized and must be reconstituted with diluent and homogenized at the time of application. The lyophilised vaccine is presented as a white powder and the sterile diluent is translucent. Both are presented in vial of colorless neutral glass.
  Arms: MenCC-BIO Vaccine
Biological: Combined - CRM197 — The comparison is against meningococcal C vaccine produced by the Foundation Ezequiel Dias (FUNED), licensed by ANVISA and currently provided by the National Immunization Program in the child's immunization schedule. This vaccine containing 10 microgram of meningococcal C oligosaccharide conjugate 12,5-25microgram of CRM197 protein of Corynebacterium diphtheriae, and presents aluminum hydroxide (0.3 to 0.4 milligram Al3 +) in its formulation. It is also a lyophilized product must be reconstituted and homogenized before use. The meningococcal C vaccine adsorbed (combined - CRM197) comprises two frascos- ampoule, containing a white or off-white lyophilized powder and another vial containing a white opalescent suspension (diluent).
  Arms: combined - CRM197

SUMMARY:
TYPE / DESIGN STUDY: Clinical trial phase II / III, randomized, double-blind, national multi-center, with a total of 1,644 research participants stratified into 3 groups according to age for starting of the primary vaccination schedule (Stratum I - 11 to 19 years, Stratum II - 1 to 10 years; Stratum III - less than 1 year old).

BACKGROUND / STUDY CASE: Clinical trial phase II / III, which purpose is to evaluate immunogenicity, safety and reactogenicity of the vaccine against meningococcus C, conjugated to tetanus toxoid, developed by Bio-Manguinhos / FIOCRUZ (MenCC-Bio). The hypothesis of the study is that MenCC-BIO vaccine is safe and not inferior in terms of immunogenicity to the comparator vaccine currently available for the National Immunization Program in the child's immunization schedule. Thus, MenCC-Bio vaccine may meet the need for expansion of the target age group of vaccination in routine public health services and will be available to the National Immunization Program as a strategy to ensure sustainability and self-sufficiency to vaccination policy.

OBJECTIVES PRIMARY: To assess the immunogenicity of MenCC Bio-vaccine in patients from 3 months to 19 years of age, in relation to the vaccine against meningococcus C currently provided by the National Immunization Program. To evaluate the safety and reactogenicity of MenCC Bio-vaccine in patients from 3 months to 19 years old.

SECONDARY OBJECTIVES: Evaluate the cellular immune component to meningococcal C conjugate vaccine in a subset of survey participants, aged 11 to 19 years.

STUDY POPULATION: Individuals of both sexes, healthy, aged between 3 months and 19 years, attending the campus of Fiocruz / Rio de Janeiro, or municipal health units in Rio de Janeiro (living in areas covered by the municipal units health participants) that fit in the study eligibility criteria.

NUMBER OF CENTRES: Two Clinical sites.

STUDY DURATION: Estimate of 19 months.

INTERVENTION / TREATMENT: Two intervention groups (MenCC-BIO Vaccine and Comparator) in three age groups, with specific vaccination schedules. For the age groups I and II are applied 2 doses ideal interval of 6 months between them. In stratum III, are recommended 3 doses of the vaccine, at ages 3, 5 and 12 months of age, according to calendar of the National Immunization Program.

OUTCOMES PRIMARY:

Immunogenicity:

Proportion of seroconversion defined by the seronegative status change (titles of bactericidal antibodies in children rabbit complement than 1: 8) to seropositive (titers of bactericidal antibodies in larger rabbit complement or equal to 1: 8) or increase 4 times of post vaccinal compared to pre-vacianais after the full vaccination schedule by age stratum.

Geometric mean antibody titers (TGM) pre- and post-vaccination, for each vaccine group, and the ratio of these securities after the full vaccination schedule by age stratum.

Safety and reactogenicity: Frequency and intensity of adverse events solicited and unsolicited, which occurred 30 days after vaccination.

SECONDARY OUTCOME : cell detection B (CD19 +) memory phenotype (CD27 + IgD +, CD27 + IgD) in a subgroup of patients in the age stratum I (11-19 years old). ADDITIONAL INFORMATION age escalation, with interim analysis of inter-layer security and approval by the Security Independent Monitoring Committee of progression to the next lower age stratum.

DETAILED DESCRIPTION:
Status: Not yet recruiting: participants are not yet being recruited.

ELIGIBILITY:
Inclusion Criteria:

* Be current on the national calendar own vaccination for the age group (except for meningitis C vaccine - see exclusion criteria).
* Available for monitoring throughout the study period.
* Willing to provide name, address, telephone number and other information so that we can contact the person if necessary (eg in case of missing the scheduled visit).
* Willing to strictly follow the study protocol.
* Legal Responsible and research participants with the ability to understand and sign the free and informed consent and the informed free consent term, according to the particularities of the age groups.
* Understand the impossibility to participate in another clinical trial during the time you are participating in the study.
* intellectual level or that of his legal guardian (if applicable according to age research participant) for the filling in the forms for registration of signs and symptoms at home.

Exclusion Criteria:

* Previous vaccination against meningococcus
* Personal history of meningitis of any kind.
* Personal history of anaphylaxis, asthma, urticaria or other hypersensitivity reaction to previous vaccinations or who have allergies or hypersensitivity to the study vaccine components.
* Use of allergy shots with antigens within 14 days or less prior to vaccination.
* Immunoglobulin Use in the last 12 months prior to vaccination.
* Use of blood products in the 12 months prior to vaccination.
* Use of any type of vaccine within 30 days before study vaccination.
* The use of injectable vaccines least 30 days after the vaccination study.
* Chronic use of any medication, except homeopathic medicines, medication trivial as saline nasal use and vitamins, and birth control.
* Prior use of immunosuppressant or cytotoxic medication. individuals are acceptable to have made use of this type of medication not immunosuppressant doses for over 6 months as nasal steroids for allergic rhinitis or topical steroids for uncomplicated dermatitis.
* In use of systemic treatment with high doses of steroids (for example, 1 mg / kg / day of prednisone for at least 14 days, or equivalent) or history of chronic use of high power inhaled corticosteroids (e.g., 800 ug per fluticasone day).
* Use of any type of medication in clinical trials over a period of one year prior to vaccination.
* Personal history of neurological, cardiovascular, respiratory, hepatic, renal, hematologic, rheumatic or autoimmune clinically significant (diseases that have led to hospitalization or prolonged treatment).
* Personal history of bleeding disorders diagnosed by a physician or account of capillary fragility (eg. Bruising or bleeding without justifiable cause).
* Personal history of seizures.
* personal history of psychiatric disease that hinders adherence to protocol, such as psychosis, obsessive-compulsive neuroses, bipolar disorder being treated, diseases that require treatment with lithium and suicidal ideas in the past 5 years prior to enrollment.
* Personal history of active malignant disease (eg any type of cancer) or treated you can use during the study.
* Personal history of sickle cell anemia.
* Asplenia (absence of spleen or removal thereof).
* HIV positive or history of any immunosuppressive disease.
* Pregnancy or breastfeeding. Additional criteria for female participants of childbearing age: negative pregnancy test prior to application of doses of vaccines.
* The presence of any disorder that, in the opinion of the principal investigator, may interfere with the evaluation of the study objectives.
* Inability to collect blood for evaluation of pre-vaccine based (baseline).

Ages: 3 Months to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1644 (Estimated)
Dates: Start 2018-09-25 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Measure seroconversion proportion | Immediately before administration of the booster dose
Measure geometric mean antibody titers (TGM) | Immediately before administration of the booster dose
Measure frequency and intensity of adverse events solicited and unsolicited | 30 days after vaccination
Measure seroconversion proportion | 30 days after administration of the booster dose
Measure the ratio of antibody titers | 30 days after administration of the booster dose
Measure the ratio antibody titers | Immediately before administration of the booster dose
Measure geometric mean antibody titers (TGM) | 30 days after administration of the booster dose

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana de Noronha, Doc, Principal Investigator — The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz)
Locations (1):
- • Unidade de Ensaios Clínicos para Imunobiológicos/Instituto de Tecnologia em Imunobiológicos de Bio-Manguinhos/Fiocruz, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No